CLINICAL TRIAL: NCT07191730
Title: Machine Learning Score Prediction of Cardiotoxicity in Cancer Patients Receiving Anthracycline Chemotherapy or HER-2-Targeted Therapies
Brief Title: ML Score Prediction of Cardiotoxicity in Cancer Patients Receiving Anthracycline Chemotherapy or HER2-Targeted Therapies
Acronym: ML-CardioTox
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: 23-0270
Record Dates: First submitted 2025-08-25; First posted 2025-09-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-08

CONDITIONS: Cardiotoxicity; Heart Failure; Neoplasms; Breast Neoplasms
Keywords: Cancer Therapy-Related Cardiac Dysfunction; Anthracyclines; HER2-targeted Therapy; Cardio-Oncology; Machine Learning
MeSH Terms: conditions — Cardiotoxicity; Heart Failure; Neoplasms; Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Cancer treatments have improved substantially over the past decades, but some effective therapies such as anthracyclines and HER2-targeted agents are associated with severe cardiovascular adverse effects, including heart failure. Existing cardiovascular risk prediction scores have limited evidence in this setting.

The ML-CardioTox study is a prospective, multicenter, observational cohort conducted in 15 centers in France. The primary objective is to develop a one-year prediction score for cancer therapy-related cardiotoxicity using machine learning methods. A dedicated software platform will be used to standardize data collection and support integration of artificial intelligence tools.

A total of 600 patients treated with anthracyclines or HER2-targeted therapies in cardio-oncology clinics will be enrolled over a one-year inclusion period starting in December 2024, with a 12-month follow-up. The primary endpoint is the occurrence of cardiotoxicity as defined by the 2022 European Society of Cardiology guidelines (hospitalization for heart failure, initiation or escalation of diuretic therapy, decline in cardiac function on imaging, or increase in cardiac biomarkers such as troponin or natriuretic peptides).

Secondary objectives include comparison of the predictive performance of the machine learning-derived score with the established HFA-ICOS risk score. Patients will be managed according to routine clinical practice.

This study aims to improve prognostic stratification tools for patients receiving anthracyclines or HER2-targeted therapies, with the goal of better identifying those at high risk of developing cardiotoxicity during follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Planned follow-up in cardio-oncology clinic as part of a baseline pre-treatment evaluation before a sequence of anthracycline and/or HER2-targeted therapy, according to the 2022 ESC recommendations
* Inclusion regardless of prior exposure to potentially cardiotoxic anticancer therapies or thoracic radiotherapy

Exclusion Criteria:

* Patients not covered by the French national health insurance system (Sécurité Sociale)
* Patients for whom 12-month follow-up is planned outside the center performing the baseline pre-treatment evaluation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with cancer scheduled to receive anthracyclines and/or HER2-targeted therapy, referred to cardio-oncology clinics in 15 participating French centers for a baseline pre-treatment evaluation and planned follow-up. Consecutive eligible patients will be enrolled over a 12-month inclusion period, with a 12-month follow-up.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2027-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Incidence of cardiotoxicity at 12 months | 12 months after initiation of anthracycline or HER2-targeted therapy.
  Cardiotoxicity defined as a composite outcome, according to the 2022 ESC guidelines: hospitalization for heart failure OR initiation or escalation of diuretic therapy for signs or symptoms of heart failure OR decrease in left ventricular ejection fraction (LVEF) by >10 percentage points from baseline or to a value <40% OR relative decrease in global longitudinal strain (GLS) ≥15% from baseline OR new increase in cardiac biomarkers (troponin or NT-proBNP/BNP). Events will be adjudicated by an independent committee.

SECONDARY OUTCOMES:
Predictive performance of machine learning-derived cardiotoxicity risk score | 12 months after initiation of anthracycline or HER2-targeted therapy.
  Performance assessed by AUC-ROC, AUC-PR, balanced accuracy, F1 score, PPV, NPV, McNemar's test, and Brier score. Unit of Measure: AUC values, accuracy (%), predictive values (%).
Comparison of predictive performance with HFA-ICOS risk score and traditional Cox model | 12 months after initiation of anthracycline or HER2-targeted therapy.
  Direct comparison of ML-derived risk score vs. HFA-ICOS and Cox model. Unit of Measure: Difference in AUC values (%), statistical comparison (DeLong test).
Correlation between baseline prognostic factors and cardiotoxicity at 12 months | 12 months after initiation of anthracycline or HER2-targeted therapy.
  Evaluation of demographic, clinical, biological (including biomarkers), and echocardiographic factors for correlation with cardiotoxicity occurrence. Unit of Measure: Odds ratios (OR) or hazard ratios (HR) with 95% confidence intervals.